CLINICAL TRIAL: NCT05058690
Title: Artificial Intelligence to Improve Cardiometabolic Risk Evaluation Using CT Scans
Acronym: ACRE-CT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caristo Diagnostics Limited (Industry)
Collaborators: University of Oxford (Other); University of Leeds (Other); Milton Keynes University Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ACRE-CT
Record Dates: First submitted 2021-09-08; First posted 2021-09-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pre-diabetes; Diabetes Mellitus
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — Glucose Tolerance Test

STUDY DESIGN:
Intervention Model Description: Multi-centre, prospective cohort, study
Who Masked: Participant
Masking Description: Personal identifiable data (including the code-break/participant key) collected at the recruitment site will be recorded electronically on a database that is stored on an access-restricted computer and either encrypted and/or located on a secure server and accessed only by authorised staff. Any copies leaving the study site will be completely anonymised/de-identified. Informed consent forms that contain participant names will be stored securely at study sites in locked cupboards and will only be accessible to study staff and authorised personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals who had a CCTA as part of their clinical care (Experimental): Approximately 90 individuals who had a CCTA as part of their clinical care (45 identified as having an abnormal FatHealth algorithm calculation and 45 with a normal FatHealth algorithm calculation) will undergo OGTT which is evaluable;
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test
- Individuals who had a chest CT as part of their clinical care (Experimental): Approximately 90 individuals who had a chest CT as part of their clinical care (45 identified as having an abnormal FatHealth algorithm calculation and 45 with a normal FatHealth algorithm calculation) will undergo OGTT which is evaluable.
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — * Obtain blood sample for glucose assessment (time "0" sample). This may be obtained via venepuncture or after cannula insertion.
  * Test a small sample using a near patient glucose testing meter. If the result on the glucose meter is greater than or equal to 11mmol/L, send the blood sample urgently to lab. If it is confirmed by biochemistry to be above 11mmol/L, there is no need to continue test.
  * If the result is less than 11mmol/L on meter, give the patient the glucose solution to drink.
  * Collect a further blood sample at 120 minutes.
  * Send samples all together to laboratory for glucose measurement.

SUMMARY:
To validate the ability of the FatHealth algorithm to identify individuals with pre-diabetes and with type 2 diabetes mellitus

DETAILED DESCRIPTION:
This multicentre prospective study will evaluate the ability of the FatHealth technology to correctly identify individuals with pre-diabetes and diabetes, validating the technology against the current gold-standard diagnostic method, oral glucose tolerance testing.

Participants will be individuals who have undergone a CT scan of the chest (coronary CT angiogram [CCTA] or CT chest) as part of observational cohort studies.

Participants will be invited for an oral glucose tolerance test (OGTT), which is the current gold-standard method for detecting pre-diabetes and diabetes mellitus. All patients must have an evaluable OGTT. The study population will include:

1. Approximately 90 individuals who had a CCTA as part of their clinical care (45 identified as having an abnormal FatHealth algorithm calculation and 45 with a normal FatHealth algorithm calculation) will undergo OGTT which is evaluable; and
2. Approximately 90 individuals who had a chest CT as part of their clinical care (45 identified as having an abnormal FatHealth algorithm calculation and 45 with a normal FatHealth algorithm calculation) will undergo OGTT which is evaluable.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study. Male or Female, aged 18 to 80 years.
* Body mass index (BMI) ≥ 25kg/m2
* FatHealth status assessed as the following:

  * Elevated FatHealth status (50% of participants)
  * Non-elevated FatHealth status (50% of participants)

Exclusion Criteria:

* Participant is unable or unwilling to give informed consent
* Participant is unable to understand English language
* Confirmed diagnosis of diabetes mellitus treated with oral medication or Insulin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants identified with pre-diabetes/type 2 diabetes mellitus when fasting blood sample test results are compared against FatHealth algorithm results | Baseline
  The investigators will measure if the fasting blood sample results indicate that the individual has pre-diabetes/type 2 diabetes mellitus and compare if our FatHealth algorithm indicates the same results for the individual

SECONDARY OUTCOMES:
Number of participants identified with pre-diabetes/type 2 diabetes mellitus when oral glucose tolerance test results are compared against FatHealth algorithm results | 120 minutes after baseline
  The investigators will measure if the oral glucose tolerance test results indicate that the individual has pre-diabetes/type 2 diabetes mellitus and compare if our FatHealth algorithm indicates the same results for the individual

IPD SHARING:
Plan to Share IPD: No
No plans to share participant data with other researchers